CLINICAL TRIAL: NCT07203222
Title: Comparison of the Efficacy of Low-Dose Laser and Transcutaneous Electrical Nerve Stimulation in Subacute Hemiplegic Shoulder Pain, and the Effect of Treatments on Upper Extremity Function and Quality of Life
Brief Title: Comparison of Effectiveness of Low Dose Laser and Transcutaneous Electrical Stimulation in Hemiplegic Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-066
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: Hemiplegic shoulder pain; Low Dose Laser; TENS; Ultrasonographic evaluation; Upper extremity function; stroke
MeSH Terms: conditions — Stroke | interventions — Lasers; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose Laser Group (Experimental): Patients who will undergo low laser therapy
  Interventions: Device: Low Dose Laser; Other: Conventional physical therapy
- TENS group (Active Comparator): Patients who will undergo TENS therapy
  Interventions: Device: TENS; Other: Conventional physical therapy
- Conventional Therapy (Active Comparator): Patients who will undergo conventional therapy
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Low Dose Laser — Patients with subacromial-subdeltoid bursa, m. deltoideus, m. biceps longus, m. infraspinatus, and m. supraspinatus muscles (at the most painful point of the muscles) with a 13-diode Gallium-Aluminium-Arsenide laser device (Intelect Mobile Laser) with a wavelength of 850 nm and 50 mW, 4 Joules per day, 20 seconds, for a total of 15 laser sessions.
  Arms: Low Dose Laser Group
Device: TENS — TENS therapy will be administered using the TENS device (Intelect Advanced Therapy System) for a total of 15 sessions, 5 days a week, 20 minutes per day, at a dose of 20-40 mA.
  Arms: TENS group
Other: Conventional physical therapy — Only conventional physiotherapy is planned to be administered to patients.

SUMMARY:
The primary aim of this study is to compare the efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) and Low Level Laser Therapy (LLLT), which are analgesic modalities that play an important role in the treatment of this frequently encountered complication. The secondary aim of the study is to evaluate its effectiveness on upper extremity function, quality of life, sleep, and fatigue.

DETAILED DESCRIPTION:
Stroke is a leading cause of morbidity and mortality worldwide. (1) Hemiplegic shoulder pain (HSP) is one of the common complications seen in up to 40% of stroke patients and negatively affects the rehabilitation process. (2) It is also a significant complication that prolongs hospital stay. Therefore, developing effective treatment strategies is extremely important.

The primary aim of our study is to compare the efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) and Low Level Laser Therapy (LLLT), which are analgesic modalities that play an important role in the treatment of this frequently encountered complication.

Treatment methods used for hemiplegic shoulder pain: Exercises (joint range of motion, stretching and strengthening exercises), physical therapy agents, kinesiology taping, transcutaneous electrical nerve stimulation (TENS), suprascapular nerve block (SSNB), suprascapular nerve pulsed radiofrequency (PRF), botulinum toxin type A (BoNT-A) intramuscular injections, corticosteroid injections, segmental neuromyotherapy (SNMT), trigger point dry needling (TrPs-DN), robot-assisted shoulder rehabilitation therapy (RSRT), platelet-rich plasma (PrP) injection, repetitive transcranial magnetic stimulation ( rTMS), peripheral nerve stimulation (PNS), neuromuscular electrical stimulation (NMES), functional electrical stimulation (FES), and interferential current stimulation (IFC) play a role in the management of the hemiplegic shoulder pain clinic. (3)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years
* Patients with shoulder pain on the hemiplegic side *Mini mental state examination ≥ 25
* History of stroke within the last 2 weeks to 6 months
* Patients with shoulder pain scoring 40-100 points on the visual analogue scale (moderate to severe) will be included.

Exclusion Criteria:

* Patients who refuse to provide written consent or attend follow-up visits
* Being under 18 years of age
* Patients with motor aphasia
* Patients who have had a shoulder injection within the last 3 months
* Patients who have undergone upper extremity botulinum toxin application within the last 6 months

  *Pregnant women or those planning to become pregnant
* Inflammatory rheumatic disease
* Patients who have undergone shoulder injury and surgery prior to stroke
* Patients with other conditions that could explain shoulder pain
* Patients with complex regional pain syndrome
* Patients with a history of epilepsy, pacemaker, or arrhythmia diagnosis
* Malignancy
* Diseases such as Alzheimer's or dementia that cause cognitive impairment -History of psychiatric disorders such as major depression or personality disorders
* Alcohol and drug addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
  It is a method used to measure a person's level of pain or discomfort. The VAS allows patients to quantitatively express their level of pain or discomfort based on their own perceptions. The VAS is scored on a scale of 0-100.
  Mild: 10-39, Moderate: 40-79, Severe: 80-100

SECONDARY OUTCOMES:
Modify Ashworth Scale | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
  It is the most commonly used assessment method for spasticity on an international platform. The joint should be moved passively, repeatedly and rapidly, and resistance should be graded according to the examination findings. It is graded as 0, 1, 1+, 2, 3, 4.
Fugl Meyer Upper Extremity Motor Function Scale | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
  It is a scale used to assess sensorimotor impairment in patients with a history of stroke. It is designed to evaluate motor function, balance, sensation, and joint function in patients with hemiplegia. Each task is scored on a scale of 0 to 2. The total score ranges from 0 to 66.
Joint Range of Motion (ROM) Measurement | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Stroke-Specific Quality of Life Scale | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Barthel Index | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Beck Depression Scale | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Caregiver Burden Scale | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Fatigue assessment scale | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Pittsburgh Sleep Quality Index | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
Ultrasonographic findings | patients will be checked on first day of hospitalization, after treatment at 4 weeks and after treatment 3 months
  Sonographic criteria have been defined based on previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: nihal tezel, associate professor, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes